CLINICAL TRIAL: NCT00895986
Title: Achieving and Maintaining Glycemic Control: Using Conversation Maps to Reinforce Self-Care
Brief Title: Using Conversation Maps to Reinforce Self-Care
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Joslin Diabetes Center (Other)
Collaborators: American Diabetes Association (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: ADA 7-08-CR-62; CHS #08-07
Record Dates: First submitted 2009-05-07; First posted 2009-05-11 (Estimated); Last update posted 2012-10-18 (Estimated); Status verified 2012-10

CONDITIONS: Type 2 Diabetes
Keywords: Diabetes; Education
MeSH Terms: conditions — Diabetes Mellitus, Type 2; Diabetes Mellitus

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- 1 (Experimental): Conversation Maps Diabetes Education
  Interventions: Behavioral: Conversation Maps Diabetes Education
- 2 (Experimental): Heart Healthy Living Diabetes Education
  Interventions: Behavioral: Heart Healthy Living Diabetes Education

INTERVENTIONS:
Behavioral: Conversation Maps Diabetes Education — The Conversation Maps program is a set of innovative, interactive diabetes education tools developed by the Healthy Interactions, Inc (Healthy I) and endorsed by the American Diabetes Association. It consists of four conversation maps covering: 1) Diabetes Overview, 2) Diabetes and Healthy Eating, 3) Blood Glucose and Monitoring, and 4) The Natural Course of Diabetes (a fifth map covering gestational diabetes will not be used in this study), and a program manual to help educators successfully implement the program.
  Arms: 1
Behavioral: Heart Healthy Living Diabetes Education — The Joslin Clinic offers a series of two 120-minute classes specifically for people with diabetes that address dyslipidemia and blood pressure problems. A registered nurse and/or a registered dietitian teach the classes, which have a formal written curriculum, including PowerPoint slides.
  Arms: 2

SUMMARY:
Many people with type 2 diabetes are not able to keep their blood glucose in good control. Improving blood glucose control and maintaining that improvement is important for diabetes patients because doing so delays the onset and progression of severe complications of diabetes. Although educational programs may be helpful, their effect is not always long-lasting. This project is studying whether the Conversation Maps program (an interactive diabetes education program) reinforces diabetes education and information and thus helps type 2 diabetes patients take better care of their diabetes and blood glucose levels. Half of the patients will attend the Conversation Maps program and half of the patients will attend an educational program about blood pressure and cholesterol. Also, all patients will come in for 4 or 5 appointments to complete surveys and other tests and have their blood drawn. The group of patients who attend the Conversation Maps program will be compared to the group of patients who attend the blood pressure and cholesterol program to see if the educational programs helped diabetes patients to improve their diabetes control and quality of life and to maintain that improvement over time.

ELIGIBILITY:
Inclusion Criteria:

* Ages 25-75 years
* Diagnosis of type 2 diabetes mellitus
* Two A1c levels ≥7.0 % (above ADA target)
* 2 years since initial diagnosis. This will provide a minimum of two-years experience with diabetes treatment. Also, excluding those who are newly diagnosed will prevent improvement due to newly prescribed medications from confounding study results.
* Attended one of Joslin's group education programs or comparable 3-hour (or more) educational programs and/or appointments

Exclusion Criteria:

* Severe complications of diabetes including renal disease (microalbumin >300 ug/mg), severe peripheral diabetic neuropathy and/or severe peripheral vascular disease, symptomatic severe autonomic neuropathy, that may place participants at risk when increasing activity levels.
* Proliferative diabetic retinopathy based on dilated eye examination within one year of study entry. Patients whose eye disease is successfully treated will be included.
* Current or planned pregnancy
* A1c levels less than 7.0% (normal range 4.0 - 6.0%) and A1c levels greater than 14%.
* A history of severe, unstable myocardial infarction, congestive heart failure or other severe cardiac disease, or severe hypertension (systolic ≥160 mmHg or diastolic ≥ 90 mmHg) (increased risk when mildly increasing physical activity).
* A diagnosis of bipolar disorder, schizophrenia, mental retardation, organic mental disorder, and alcohol or drug abuse will be excluded, as well as patients currently undergoing psychiatric treatment. These exclusions are being made to avoid confounds due to concurrent changes in mental status and the effects of ongoing psychiatric treatment.
* Used Conversation Maps as an educational tool
* Started a new diabetes medication (pills or insulin) in past three months

Ages: 25 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 134 (Actual)
Dates: Start 2008-12; Primary Completion 2012-03 (Actual); Study Completion 2012-03 (Actual)

PRIMARY OUTCOMES:
Improved frequency of recommended self-care behaviors (Self-Care Inventory-R) | 3, 6, and 12 months post intervention

SECONDARY OUTCOMES:
HbA1c | 3, 6, and 12 months post intervention
Diabetes Quality of Life (scale) | 3, 6, and 12 months post intervention
Major mediating/moderating variables include Problem Areas in Diabetes, Brief Symptom Inventory, Coping Styles, and Confidence in Diabetes | 3, 6, and 12 months post intervention

CONTACTS AND LOCATIONS:
Overall Officials: Katie Weinger, EdD, RN, Principal Investigator — Joslin Diabetes Center
Locations (1):
- Joslin Diabetes Center, Boston, Massachusetts, United States